CLINICAL TRIAL: NCT01310790
Title: Strategy of Early Improvement of Tissue Oxygenation Decrease the Mortality of Severe Sepsis
Brief Title: Strategy of Early Improvement of Tissue Oxygenation Decrease the Mortality of Severe Sepsis and Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Septic Shock Network (Network)
Responsible Party: DaweiLIU, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSSN-6091-DaweiLiu
Record Dates: First submitted 2011-02-08; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Shock, Septic
Keywords: septic shock; lactic acid clearance; ScVO2
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: lactate group:lactate acide clearance directed group; ScvO2 group:ScvO2 directed group;control group — Patients assigned to lactate group started with the resuscitation to achieve a CVP of 8 to 12 mmHg and MAP 65 to 90 mmHg. Then if ScvO2 was less than 70 percent, red cells were transfused to achieve a hematocrit of at least 30 percent. After the CVP, MAP, and hematocrit achieved the goals, dobutamine was given until the ScvO2 was 70 percent or higher. Arterial blood lactate concentration was obtained at 6 hours and try to achieve lactate clearance was >30%.
  Patients in the ScvO2 group received the treatment as ScvO2 directed therapy protocol for at least 6 hours and maintained for 72 hours. The protocol was the same as that of lactated directed therapy with the exception of blood lactate concentration testing.
  Patients in the control group received the treatment as the same protocol for maintaining CVP and MAP in that of lactated directed therapy. ScvO2 and arterial blood lactated concentration were not necessary to obtain.

SUMMARY:
The impact of lactate guided therapy on septic shock has not been extensively investigated, however the goal directed therapy has been used for years. The investigators aim was to test the hypothesis that lactate directed hemodynamic therapy is associated with improving the outcome of patients with septic shock by comparing different goal directed strategies which have been commonly recommended clinically.

In this multicenter, randomized trial, the investigators assigned patients with septic shock to three groups: Patients were treated with hemodynamic therapy directed either by conventional parameters treatment (control group), or central venous oxygen saturation (ScvO2), or blood lactate respectively in each group. The primary outcome was the rate of death at 28 days after randomization and in-hospital mortality; secondary end points include hemodynamic states, time to goal-achievement.

DETAILED DESCRIPTION:
This prospective, randomized, controlled and multi-center study was performed in 6 closed intensive care units (ICU) of academic tertiary hospitals. Adult patients with septic shock admitted to the hospitals from 2005 to 2008 were assigned to the study eligibility. Eligible patients were centrally randomized using sealed envelopes into one of the three groups which included lactate, ScvO2, and control groups. The criteria of septic shock included two of four criteria for the systemic inflammatory response syndrome and systolic blood pressure lower than 90 mmHg or decrease of systolic blood pressure more than 40 mmHg after fluid challenge and the clinical signs of tissue hypoperfusion, including oliguria, blood lactate concentration of 4 mmol/L or more and consciousness alteration. The patients were excluded if they meet any one of follows: an age of less than 18 years, pregnancy, an acute cerebral vascular event (Glasgow coma score < 5), acute myocardial infarction or acute coronary syndrome, massive pulmonary embolism, status asthmaticus, a primary diagnosed cardiac dysrhythmias, contraindication to central venous catheterization, active gastrointestinal hemorrhage, massive intraabdominal infective focus without drainage, severe bronchopleural fistula, seizure, during chemotherapy or immunosuppressive therapy, or end stage of the diseases.

The protocol was approved by Institutional Ethics Committee. The informed consents were obtained from all patients or their legally authorized next of kin. The patients or their legal surrogate decision makers were informed of their right to refuse the study procedures at any time during the protocols were performed.

The case report forms (CRF) were sent to each site from the principal investigator with the protocols, which were randomly sealed in a serial of envelopes. After patients' enrollment, the CRFs were filled by the attending physicians at each site according to the protocol of each group. End points were 28-day mortality and in-hospital mortality until 90 days. The demographic data, acute physiological and chronic evaluation score (APACHE) II and other data from patients' basic condition were recorded at enrollment day. The protocol related data were collected at baseline and each hour for 6 hours and then at 12, 24, 36, 48, 60, 72 hours. The ICU and hospital length of stay were also noted and patients were followed up to day 28 and discharge from hospital for mortality. The protocol implementation and data collection stopped when patients or their families wished to withdraw from the program or refuse further treatment or a patient's death.

ELIGIBILITY:
Inclusion Criteria:

* severe sepsis and septic shock patients

Exclusion Criteria:

* <18 years old;
* pregnant woman;
* AMI;
* cerebral hemorrhage;
* contraindication for S-G catheter
* Brainstem death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
mortality | in-hospital
  Because some patients stayed in hospital for a quite long time,so when we made statistics,we defined that if the patient still alive after involved 90 days, this patient was in-hospital lived.

CONTACTS AND LOCATIONS:
Overall Officials: Dawei Liu, M.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Critical Care Department, Peking Union Medical Hospital, Beijing, China